CLINICAL TRIAL: NCT04137536
Title: Phase Ib Treatment of Advanced Pancreatic Cancer With Anti-CD3 x Anti-EGFR-Bispecific Antibody Armed Activated T-Cells (BATs)
Brief Title: A Study of Armed, Activated T-Cells in Patients With Advanced Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-463
Record Dates: First submitted 2019-10-21; First posted 2019-10-24 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Pancreatic Cancer; Advanced Pancreatic Cancer; Pancreatic Adenocarcinoma; Pancreatic Neoplasms
Keywords: EGFR-BAT; bispecific antibody-armed activated T cells; Pancreatic cancer; memorial sloan kettering cancer center; 18-463
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pancreatic Adenocarcinoma (Experimental): Participants have metastatic pancreatic cancer who have received at least first line chemotherapy and have disease progression during or within 6 months of treatment.
  Interventions: Drug: anti-EGFR-bispecific antibody armed activated T-cells

INTERVENTIONS:
Drug: anti-EGFR-bispecific antibody armed activated T-cells — Phase I:
  * First 3 participants, twice weekly infusions of 10^10 EGFR BATs infusions
  * If there is toxicity in 0 or 1 of 3 participants, 3 additional participants will be added to the dose level of up to 10^10.
  * If >/= 2 of 6 participants experience DLTs, then the dose will be reduced to 7.5 x 10^9 per infusion
  * If only 0 or 1 participants has toxicity in the first 6, then the study will proceed to enroll in the expansion cohort
  Expansion cohort:
  - 8 infusions of 7.5 x 10^9 or 10^10 EGFR BATs in 22 evaluable participants (including the 6 participants treated at the maximum tolerated dose in Phase I)
  Other Names: EGFR BATs

SUMMARY:
The purpose of this study is to find the safest dose and identify any bad side effects of EGFR-BATs (bispecific antibody-armed activated T cells) for people with advanced pancreatic cancer who have already received first-line standard chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological proof of pancreatic adenocarcinoma. Must have metastatic pancreatic cancer who have received at least first line chemotherapy. Disease stability or progression during or within 6 months after treatment with 5-Fluorouracil (5-FU)- or gemcitabine-based chemotherapy. KPS>/= 70% or SWOG performance Status 0 or 1
* Evaluable disease by iRECIST criteria
* Absolute Neutrophil Count (ANC) >/= 1,000/mm^3
* Lymphocyte count >/= 400/mm^3
* Platelet Count >/= 75,000/mm^3
* Hemoglobin >/= 8 g/dL
* Serum Creatinine < 2.0 mg/dl, Creatinine Clearance >/=50 ml/mm (can be calculated or measured)
* Total Bilirubin </= 2 mg/dl (biliary stent is allowed)
* SGPT and SGOT <5.0 times normal
* LVEF >/= 55% at rest (<UGA or Echo)
* Age >/= 18 years at the time of consent (Written informed consent and HIPAA authorization for release of personal health information)
* Females of childbearing potential, and males, must be willing to use an effective method of contraception
* Females of childbearing potential must have a negative pregnancy test within 7 days of being registered for protocol therapy

Exclusion Criteria:

* Any chemotherapy related toxicities from prior treatment, > grade 2 per CTCAE v4.0
* Known hypersensitivity to cetuximab or other EGFR antibody
* Treatment with any investigational agent within 14 days prior to being registered for protocol therapy
* Symptomatic brain metastasis
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. Steroid premedication for imaging scans is allowed. Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Serious non-healing wound, ulcer, bone fracture, major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to being registered for protocol therapy
* Active liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis
* Known HIV infection
* Active bleeding or a pathological condition that is associated with a high risk of bleeding (therapeutic anticoagulation is allowed)
* Has an active infection requiring systemic therapy
* A serious uncontrolled medical disorder that in the opinion of the Investigator may be jeopardized by the treatment with protocol therapy.
* Females must not be breastfeeding
* Patient may be excluded if, in the opinion of the PI and investigator team, the patient is not capable of being compliant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Evaluate toxicity | 1 year
  The NCI CTEP CTCAE v4.0 will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Yu, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Virginia (Specimen Analysis), Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- [Derived] Park JA, Santich BH, Xu H, Lum LG, Cheung NV. Potent ex vivo armed T cells using recombinant bispecific antibodies for adoptive immunotherapy with reduced cytokine release. J Immunother Cancer. 2021 May;9(5):e002222. doi: 10.1136/jitc-2020-002222. PMID 33986124
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org